CLINICAL TRIAL: NCT03907852
Title: A Phase 1/2 Single Arm Open-Label Clinical Trial of Gavocabtagene Autoleucel (Gavo-cel) in Patients With Advanced Mesothelin-Expressing Cancer
Brief Title: Phase 1/2 Trial of Gavo-cel (TC-210) in Patients With Advanced Mesothelin-Expressing Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TCR2 Therapeutics (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCR2-18-01
Record Dates: First submitted 2019-04-01; First posted 2019-04-09 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Mesothelioma; Mesothelioma, Malignant; Mesothelioma; Pleura; Mesotheliomas Pleural; Mesothelioma Peritoneum; Cholangiocarcinoma; Cholangiocarcinoma Recurrent; Ovarian Cancer; Non Small Cell Lung Cancer; Non Small Cell Lung Cancer Metastatic; High Grade Ovarian Serous Adenocarcinoma
MeSH Terms: conditions — Mesothelioma; Mesothelioma, Malignant; Cholangiocarcinoma; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — fludarabine; Cyclophosphamide; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lymphodepletion followed by gavo-cel (Experimental): fludarabine 30 mg/m2/d on days -7 through -4 and cyclophosphamide 600 mg/m2/d on days -6 through -4 followed by gavo-cel
  Interventions: Biological: gavo-cel; Drug: fludarabine; Drug: cyclophosphamide
- Lymphodepletion followed by gavo-cel plus nivolumab (Experimental): fludarabine 30 mg/m2/d on days -7 through -4 and cyclophosphamide 600 mg/m2/d on days -6 through -4 followed by gavo-cel with nivolumab 360mg every 3 weeks starting on Day 21 post gavo-cel
  Interventions: Biological: gavo-cel; Drug: fludarabine; Drug: cyclophosphamide; Drug: Nivolumab
- Lymphodepletion followed by gavo-cel plus nivolumab and ipilimumab (Experimental): fludarabine 30 mg/m2/d on days -7 through -4 and cyclophosphamide 600 mg/m2/d on days -6 through -4 followed by gavo-cel with nivolumab 360mg every 3 weeks starting on Day 21 post gavo-cel and ipilimumab 1mg/kg every 6 weeks starting on Day 42 post gavo-cel
  Interventions: Biological: gavo-cel; Drug: fludarabine; Drug: cyclophosphamide; Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Biological: gavo-cel — gavo-cel
Drug: fludarabine — lymphodepletion chemotherapy
Drug: cyclophosphamide — lymphodepletion chemotherapy
Drug: Nivolumab — immuno-oncology agent
  Arms: Lymphodepletion followed by gavo-cel plus nivolumab; Lymphodepletion followed by gavo-cel plus nivolumab and ipilimumab
Drug: Ipilimumab — immuno-oncology agent
  Arms: Lymphodepletion followed by gavo-cel plus nivolumab and ipilimumab

SUMMARY:
Gavocabtagene autoleucel (gavo-cel; TC-210) is a novel cell therapy that consists of autologous genetically engineered T cells expressing a single-domain antibody that recognizes human Mesothelin, fused to the CD3-epsilon subunit which, upon expression, is incorporated into the endogenous T cell receptor (TCR) complex.

This Phase 1/2 study aims to establish the recommended Phase 2 dose (RP2D) and subsequently evaluate the efficacy of gavo-cel, with and without immuno-oncology agents, in patients with advanced mesothelin-expressing cancers, with overall response rate and disease control rate as the primary Phase 2 endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age at the time the Informed Consent is signed.
* Patient has a pathologically confirmed diagnosis of either Malignant Pleural/Peritoneal Mesothelioma (MPM), Serous Ovarian Adenocarcinoma, Cholangiocarcinoma, or Non-Small Cell Lung Cancer (NSCLC) at screening.
* Patient's tumor has been pathologically reviewed by the central laboratory. For Serous Ovarian Adenocarcinoma, patients must have confirmed positive MSLN expression on >/= 30% of tumor cells that are 1+, 2+, and/or 3+ by immunohistochemistry (IHC). Ovarian patients will subsequently be stratified into two groups: high MSLN expression (>/= 50% of tumor cells that are 2+ and/or 3+) or low MSLN expression (>/= 30% of tumor cells that are 1+, 2+, and/or 3+ not meeting criteria for the high MSLN expression group). MPM patients must have MSLN expression of >/= 50% of tumor cells that are 2+ and/or 3+ by IHC. Cholangiocarcinoma and NSCLC patients must have MSLN expression of >/= 30% of tumor cells that are 1+, 2+, and/or 3+ by IHC.
* Prior to gavo-cel infusion, patients must have received at least 1 systemic standard of care therapy for metastatic or unresectable disease, with the exception of Cholangiocarcinoma patients who may have elected not to pursue standard frontline therapy. Regardless of tumor type, patients must not exceed 5 prior lines of therapy (excluding bridging therapy and surgical procedures). More details provided in the clinical protocol.
* Patient has an Eastern Cooperative Oncology Group performance status 0 or 1.
* Patient has a left ventricular ejection fraction > 45% as measured by resting echocardiogram, with no clinically significant pericardial effusion.
* Patient is fit for leukapheresis and has adequate venous access for the cell collection.
* Patient must have adequate organ function as indicated by the laboratory values in the clinical protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2028-11-02 (Estimated)

PRIMARY OUTCOMES:
Phase 1- Primary Objective | DLTs within 28 days post-treatment
  Establish the recommended Phase 2 dose (RP2D) according to dose-limiting toxicity (DLT) of defined adverse events.
Phase 2- Primary Objective | ORR at 3 months; DCR based on ORR + SD lasting at least 8 weeks
  To evaluate the efficacy of autologous genetically modified T cells (gavo-cel), with or without immuno-oncology agents, in patients with MSLN-expressing unresectable, metastatic, or recurrent cancers as determined by overall response rate and disease control rate using RECIST v1.1 (or mesothelioma-specific RECIST criteria, if applicable).

CONTACTS AND LOCATIONS:
Locations (11):
- United States (10):
  - University of California, San Francisco, San Francisco, California
  - University of Miami Sylvester Cancer Center, Miami, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - National Cancer Institute, Bethesda, Maryland
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - SCRI Oncology Partners, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Hassan R, Butler M, O'Cearbhaill RE, Oh DY, Johnson M, Zikaras K, Smalley M, Ross M, Tanyi JL, Ghafoor A, Shah NN, Saboury B, Cao L, Quintas-Cardama A, Hong D. Mesothelin-targeting T cell receptor fusion construct cell therapy in refractory solid tumors: phase 1/2 trial interim results. Nat Med. 2023 Aug;29(8):2099-2109. doi: 10.1038/s41591-023-02452-y. Epub 2023 Jul 27. PMID 37501016